CLINICAL TRIAL: NCT03970317
Title: Characterization of Safety and Efficacy of Broad Band Light In Motion Treatment for Pigmented Skin Lesions on Chest, Arms and Back
Brief Title: Safety and Efficacy of Broad Band Light In Motion Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBLCIP001
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pigmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Broad Band Light (Experimental): Broad Band Light (BBL) motion treatment
  Interventions: Device: Broad Band Light

INTERVENTIONS:
Device: Broad Band Light — Broad Band Light Device
  Other Names: BBL

SUMMARY:
Evaluate safety and efficacy of Broad Band Light (BBL) motion technique treatment for pigmentation, skin tone and texture

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, 18 years or older
* Fitzpatrick skin type I-V
* Has visible signs of moderate to severe skin pigmentation
* Subject must agree to not make any changes in their skin regimen for the duration of the study, including the follow-up period
* Subject must be able to read, understand and sign Informed Consent Form
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes
* Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period
* Must be willing to adhere to the treatment and follow-up schedule and post-treatment care instructions
* Agree to not use any other procedure(s) in the treatment area during the study, such as laser- or light-based treatment, non-light based device treatment such as radiofrequency or ultrasound, injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler, chemical peel, or surgical procedure
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant or to father a child for the duration of the study

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* Any type of prior cosmetic treatment to the target area within 3 months of study participation, such as laser or light-based procedures or surgery.
* Prior injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler in the target area within 1 week of study participation.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo- pigmentation.
* Systemic use of retinoid, such as isotretinoin, or corticosteroid, as applicable, within 6 months of study participation.
* Topical use of retinoid, such as isotretinoin, corticosteroid or hydroquinone on the target area within 1 month of participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated, or unable/unlikely to refrain from tanning during the study (for example, subject's occupation requires regular sun exposure).
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Photographs | 6 weeks
  Evaluation of Photographs using Physician's Global Assessment Scale (0-4) where 0 is no change and 4 is very significant improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Refined Dermatology, Los Gatos, California, United States